CLINICAL TRIAL: NCT05767476
Title: Neurodevelopmental Outcome in Newborn With Hypoxic-ischemic Encephalopathy Treated With Therapeutic Hypothermia
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Romeo Domenico Marco, MD, PHD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3544
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Encephalopathy, Hypoxic Ischemic
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns with hypoxic-ischemic encephalopathy treated with therapeutic hypothermia
  Interventions: Diagnostic Test: Clinical and instrumental neurological assessment

INTERVENTIONS:
Diagnostic Test: Clinical and instrumental neurological assessment — Participants will be involved in serial assessment:
  * Neonatal Cranial Ultrasonography
  * Brain magnetic resonance imaging
  * Neurological assessment
  * Neurodevelopmental and cognitive assessment
  * Electroencephalogram (EEG)
  * Motor performance assessment

SUMMARY:
The goal of this observational study is to identify early signs of poor neurodevelopmental outcome by performing specific neurological, neurophysiological and neuroimaging assessments in newborns with hypoxic-ischemic encephalopathy treated with therapeutic hypothermia.

The main questions it aims to answer are:

* Identify patients at risk of neuromotor, cognitive and epileptic sequelae
* Plan early rehabilitation programs and future trials on early neuroprotection in infant at risk of neurodevelopmental disability

Participants will be involved in serial assessment:

* Before and after therapeutic hypothermia and before discharge: neurological assessment, according to the modified Sarna (t) score, Thompson's score and Hammersmith Neonatal Neurological Examination (HNNE); General Movement Assessment
* Amplitude integrated electroencephalogram (aEEG) within 6 hours of life, for 6 hours.
* Neonatal Cranial Ultrasonography within 6 hours of life, in the third and seventh day of life.
* Brain magnetic resonance imaging between 7 and 14 days.
* Electroencephalogram (EEG) within 7 days.

After discharge study population will perform:

* EEG between 3 and 6 months.
* Neurological assessment using Hammersmith Infant Neurological Examination (HINE) at 3-6-9-12 months.
* General Movement Assessment at 3 months.
* Neurodevelopmental assessment using the Griffiths Mental Development Scales at 24 months.
* Cognitive assessment using the Wechsler Preschool and Primary Scale of Intelligence between 36 and 41 months.
* Motor performance assessment using Movement ABC between 42 and 48 months.

ELIGIBILITY:
Inclusion Criteria:All infants with gestational age ≥ 35 weeks and with a body weight ≥ 1800 g were considered eligible, if they satisfied the following criteria:

* Intrapartum hypoxia defined as follows: potential of hydrogen (pH)≤ 7.0 or B.E. ≥ 16 millimole liters (mmo/L) in the 1st hour of life, obtained from cord or arterial blood, or (ii) pathological intra-partum course (e.g., abnormal foetal heart rate, cord prolapse, uterine rupture, maternal haemorrhage/trauma/epileptic seizures/cardiorespiratory arrest, shoulder dystocia, fluid meconium-stained amniotic), or Apgar score ≤5 or continuous respiratory support at 10 minutes.
* Signs of moderate or severe encephalopathy according to the Sarna (t) score and Sarna (t) staging, performed at 30-60 minutes of life: stage 2 (lethargic, poor spontaneous activity, distal flexion posture, hypotonia, weak primitive reflexes, myotic pupils, bradycardia or periodic breathing) or stage 3 (stupor/coma, decerebrate posture, spontaneous activity absent, flaccidity, primitive reflexes absent, non-reactive pupils or apnoea).
* Amplitude integrated electroencephalogram( aEEG ) by Cerebral Functional Monitoring (CFM) or electroencephalogram (EEG) for at least 30 minutes, which shows either moderate or severe electroencephalographic anomalies, or the presence of convulsions.

All enrolled infants underwent therapeutic hypothermia according to the international guideline for 72 hours.

Exclusion Criteria:

Infants with:

* gestational age <35 weeks,
* severe foetal growth restriction (body weight <1800 g),
* inability to start therapeutic hypothermia within 6 hours of birth,
* other known causes of encephalopathy (chromosomopathies, brain malformations, metabolic encephalopathies, major congenital anomalies, neonatal withdrawal syndrome), - incoercible bleeding,
* refusal of consent by the parent/guardian/legal representative

Ages: 10 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with hypoxic-ischemic encephalopathy treated with therapeutic hypotermia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 24th months
  the score in Griffiths Mental Development Scales (GMDS)

SECONDARY OUTCOMES:
Neurodevelopmental outcome | between 36th and 42th months
  the score in Wechsler Preschool and Primary Scale of Intelligence (WPPSI)
Motor coordination outcome | between 42th and 48th months.
  The score in Movement ABC (m-ABC)

CONTACTS AND LOCATIONS:
Overall Officials: Domenico M Romeo, MD,PHD, Principal Investigator — ChatolicUIT
Locations (2):
- Italy (2):
  - Domenico Marco Romeo, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli -IRRCS, Rome